CLINICAL TRIAL: NCT07143890
Title: Iron Absorption From Plant-Derived Heme Iron: An Experimental Study in Iron-Deficient Women (PHIA)
Brief Title: Iron Absorption From Plant Heme Iron
Acronym: PHIA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ETH Zurich (Other)
Responsible Party: Principal Investigator, Nicole Stoffel, Assistantprofessor, ETH Zurich
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: PHIA
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-08

CONDITIONS: Iron Deficiency (ID); Iron Absorption
Keywords: Iron sulfate; Iron fortification; plant-derived heme iron; Stable isotopes; Iron bioavailability
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (8):
- Iron chlorophyllin + Water (Experimental): 3 mg iron as Fe chlorophyllin (54Fe) + water
  Interventions: Other: Iron chlorophyllin + no-matrix
- Soy hemoglobin + Water (Experimental): 3 mg iron as soy hemoglobin (58Fe) + water
  Interventions: Other: SoyHb + no-matrix
- Ferrous sulfate + Water (negative control) (Active Comparator): 3 mg iron as ferrous sulfate (58Fe) + water
  Interventions: Other: FeSO4 + no-matrix
- Porcine hemoglobin + Water (positive control) (Active Comparator): 3 mg iron as porcine hemoglobin (57Fe) + water
  Interventions: Other: Hb + no-matrix
- Iron Chlorophyllin + Inhibitory Meal (Experimental): 3 mg iron as Fe chlorophyllin (54Fe) + maize porridge
  Interventions: Other: Iron chlorophyllin + meal-matrix
- Soy Hemoglobin + Inhibitory Meal (Experimental): 3 mg iron as soy hemoglobin (58Fe) + maize porridge
  Interventions: Other: SoyHb + meal-matrix
- Ferrous sulfate + Inhibitory Meal (negative control) (Active Comparator): 3 mg iron as ferrous sulfate (57Fe) + maize porridge
  Interventions: Other: FeSO4 + meal-matrix
- Porcine hemoglobin + Inhibitory Meal (positive control) (Active Comparator): 3 mg of iron as porcine hemoglobin (57Fe) + maize porridge
  Interventions: Other: Hb + meal-matrix

INTERVENTIONS:
Other: Iron chlorophyllin + no-matrix — Water with labelled Fe chlorophyllin (54Fe)
  Arms: Iron chlorophyllin + Water
Other: SoyHb + no-matrix — Water with labelled soy hemoglobin (58Fe)
  Arms: Soy hemoglobin + Water
Other: FeSO4 + no-matrix — Water with labelled ferrous sulfate (58Fe)
  Arms: Ferrous sulfate + Water (negative control)
Other: Hb + no-matrix — Water with labelled porcine hemoglobin (57Fe)
  Arms: Porcine hemoglobin + Water (positive control)
Other: Iron chlorophyllin + meal-matrix — Maize porridge with labelled Fe chlorophyllin (54Fe)
  Arms: Iron Chlorophyllin + Inhibitory Meal
Other: SoyHb + meal-matrix — Maize porridge with labelled soy hemoglobin (58Fe)
  Arms: Soy Hemoglobin + Inhibitory Meal
Other: FeSO4 + meal-matrix — Maize porridge with labelled ferrous sulfate (57Fe)
  Arms: Ferrous sulfate + Inhibitory Meal (negative control)
Other: Hb + meal-matrix — Maize porridge with labelled porcine hemoglobin (57Fe)
  Arms: Porcine hemoglobin + Inhibitory Meal (positive control)

SUMMARY:
Heme, an iron protoporphyin IX complex, consists of a ferrous ion captured in a porphyrin ring acting as a tetradentate ligand. The unique features of heme iron -its unusually high absorption in foods and its resistance to luminal inhibitors of iron absorption- make it a potentially interesting iron fortificant. This study aims to compare fractional iron absorption from two plant-derived heme iron compounds-iron chlorophyllin and soy hemoglobin-with ferrous sulfate (negative control) and porcine hemoglobin (positive control) in iron-deficient women. All four compounds will be intrinsically labeled with stable iron isotopes. Fractional absorption will be assessed 14 days after test meal administration via erythrocyte iron incorporation.

Absorption will be tested in two matrices: water and maize porridge (an inhibitory matrix). Each participant will consume all test conditions in a randomized order, allowing for within-subject comparisons.

ELIGIBILITY:
Inclusion Criteria:

* Serum ferritin < 45 µg/L (iron depleted)
* Body weight < 70 kg
* Body mass index 18,5 - 24,9 kg/m2 (normal weight)

Exclusion Criteria:

* Hb < 120 g/L (anemia)
* CRP > 5 µg/L (inflammation)
* Strict vegan and vegetarians
* Any metabolic, gastrointestinal kidney or chronic disease
* Consumption of mineral and vitamin supplements since screening and over the study period until last blood sample collection
* Blood transfusion over the past 6 months
* blood donation over the past 6 months
* Significant blood loss (accident, surgery) over the past 6 months
* Women who are pregnant or breast feeding
* Smoker (> 1 cigarette per week)
* Continuous/long-term use of medication (except for contraceptives)
* Therapeutic iron infusion over the past 6 months,
* Known hypersensitivity or allergy to iron supplements,
* Intention to become pregnant during the course of the studies,
* Known or suspected non-compliance, drug or alcohol abuse,
* Inability to follow the procedures of the studies, e.g. due to language problems, psychological disorders, dementia, etc. of the participant,
* Participation in another study with investigational drug within the 30 days preceding and during the present studies,
* Enrolment of the investigator, his/her family members, employees and other dependent persons

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-09-22 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Fractional Iron Absorption (%) | Day 22
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products. Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.
Fractional Iron Absorption (%) | Day 43
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products. Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.
Fractional Iron Absorption (%) | Day 64
  Fractional iron absorption will be calculated based on the shift of the iron isotope ratios in the collected blood samples after the administration of the intervention products. Fractional iron absorption will be measured as erythrocyte incorporation of the naturally occurring iron forms with different masses used to label the iron supplements.

SECONDARY OUTCOMES:
Hemoglobin (g/dL) | Day 1
  Iron status marker
Hemoglobin (g/dL) | Day 22
  Iron status marker
Hemoglobin (g/dL) | Day 43
  Iron status marker
Hemoglobin (g/dL) | Day 64
  Iron status marker
Serum Ferritin (µg/L) | Day 1
  Iron status marker
Serum Ferritin (µg/L) | Day 22
  Iron status marker
Serum Ferritin (µg/L) | Day 43
  Iron status marker
soluble Transferrin Receptor (mg/L) | Day 1
  Iron status marker
soluble Transferrin Receptor (mg/L) | Day 22
  Iron status marker
soluble Transferrin Receptor (mg/L) | Day 43
  Iron status marker
C-reactive protein (mg/L) | Day 1
  Chronic inflammation marker
C-reactive protein (mg/L) | Day 22
  Chronic inflammation marker
C-reactive protein (mg/L) | Day 43
  Chronic inflammation marker
Alpha-1-acid Glycoprotein (g/L) | Day 1
  Acute inflammation marker
Alpha-1-acid Glycoprotein (g/L) | Day 22
  Acute inflammation marker
Alpha-1-acid Glycoprotein (g/L) | Day 43
  Acute inflammation marker
Hepcidin (ng/mL) | Day 1
  A major regulator of iron absorption
Hepcidin (ng/mL) | Day 22
  A major regulator of iron absorption
Hepcidin (ng/mL) | Day 43
  A major regulator of iron absorption

CONTACTS AND LOCATIONS:
Locations (1):
- ETH Zurich, Laboratoy of Clinical Biopharmacy, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No